CLINICAL TRIAL: NCT01486784
Title: A Phase I-II Open Label Non-Randomized Study Using TL32711 for Patients With Acute Myelogenous Leukemia, Myelodysplastic Syndrome and Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 15411
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Acute Myelogenous Leukemia
Keywords: equal to or greater than age 60 years; non-M3 AML; relapsed disease; primary refractory disease; not appropriate or willing candidates for aggressive therapy; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — birinapant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase 1 DL1 (Experimental): 26mg/m2/dose IV once per week x 3 weeks of 4 week cycle
  Interventions: Drug: Birinapant
- Phase 1 DL-1 (Experimental): 17mg/m2 IV/dose once per week x 3 weeks of 4 week cycle
  Interventions: Drug: Birinapant
- Phase 1 DL-1a (Experimental): 17mg/m2/dose IV twice per week x 3 weeks of 4 week cycle
  Interventions: Drug: Birinapant
- Phase 1 DL-1b (Experimental): 17mg/m2/dose IV three times per week x 3 weeks of 4 week cycle
  Interventions: Drug: Birinapant
- Phase 1 DL-1c (Experimental): 22mg/m2/dose IV twice per week x 3 weeks of 4 week cycle
  Interventions: Drug: Birinapant
- Phase 1 DL-1d (Experimental): 17mg/m2/dose IV twice per week x 3 weeks of 4 week cycle
  Interventions: Drug: Birinapant

INTERVENTIONS:
Drug: Birinapant — IV formulation to be given weekly 3 weeks out of 4 week cycle or 4 weeks our of a 4 week cycle as a 30 minute infusion
  Other Names: TL37211

SUMMARY:
This was initially a phase I/II, open-label non-randomized study using an investigational new drug, TL32711, in patients with AML, MDS and ALL, however, the phase II portion was never initiated. This study initially targeted subjects 60 years of age and older (with non-M3 AML who have relapsed or refractory disease after standard therapy or who are newly diagnosed and subjects 18-59 (relapsed or refractory after failing 3 prior lines of therapy), and then targeted subjects 18 years of age and older with MDS and ALL.

DETAILED DESCRIPTION:
This was initially a phase I/II, open-label, non-randomized study using an investigational new drug, TL 32711, in patients with acute myelogenous leukemia. This study targeted subjects 60 years of age and older (with non-M3 AML who have relapsed or refractory disease after standard therapy or who are newly diagnosed and not candidates for standard induction therapy) and subjects 18-59 (relapsed or refractory after failing 3 prior lines of therapy). Subjects would receive the study drug in 4 weeks dosing periods via one of three different treatment schedules (once weekly, twice weekly or three times weekly dosing). They would receive treatment for up to 6 cycles, however treatment may have been extended at the discretion of the study doctor if felt to be in the best interest of the subject. Up to 46 subjects were to be enrolled on this study at the University of Pennsylvania, depending on the number of subjects needed in the Phase I component in order to determine the MTD. The primary objective of the Phase 1 component was to determine the safety and tolerability of TL32711, and the MTD in this patient population. The primary objective of the Phase 2 portion of this study was to further define the safety and tolerability, and provide preliminary efficacy data, however, the Phase II portion was never initiated.

ELIGIBILITY:
Inclusion criteria

* Subjects with a diagnosis of non-M3 AML, Relapsed or refractory ALL or Intermediate Risk 2 or High Risk disease MDS as follows:
* Subjects with a diagnosis of non-M3 AML which meets one of the following criteria:

  1. Ages 60 or older: Relapsed or refractory after at least one prior therapy for AML
  2. Ages 60 or older: Newly diagnosed in a patient with a preceding history of myelodysplastic syndrome which has been treated with azacitidine or decitabine and who are not appropriate candidates for aggressive therapy including induction followed by allogeneic stem cell transplantation
  3. Ages 18-59: Relapsed or refractory disease after failing three prior lines of therapy
* Subjects with a diagnosis of relapsed or refractory ALL: must have failed three prior lines of therapy and be 18 years of age or older.
* Subjects with a diagnosis of Intermediate Risk 2 or High Risk disease (as defined by IPSS score):

  1. Must have failed to respond/intolerant to, or progressed after a hypomethylating agent, and must not be candidates for allogeneic stem cell transplantation
  2. Life expectancy of at least 4 weeks
  3. Must have recovered from toxic effects of prior chemotherapy
  4. Patients must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing.

Exclusion criteria

* Cytotoxic chemotherapy (including azacitidine or decitabine) within the past 28 days other than hydroxyurea
* Active participation in any other investigational treatment study for AML.
* ECOG performance status greater than 2
* Uncontrolled intercurrent illness including, but not limited to: uncontrolled ongoing infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* QT interval corrected for heart rate (QTcB) greater than 480 msec (including subjects on medication). Subjects with a ventricular pacemaker for whom QT interval is not measurable may be eligible for enrollment after consultation with the drug manufacturer and study Medical Monitor, and written documentation of this approval.
* Female subjects who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 27 subjects enrolled, only 17 completed Cycle 1 of study treatment, and are therefore considered evaluable. 5 subjects withdrew or were taken off study prior to receiving study drug, 1 came off study due to disease progression, 3 were removed from the study, and 1 chose to withdraw prior to completing Cycle 1.
Period: Overall Study
Arm/Group | Phase 1 DL1 | Phase 1 DL-1 | Phase 1 DL-1a | Phase 1 DL-1b | Phase 1 DL-1c | Phase 1 DL-1d
Started | 3 | 7 | 6 | 1 | 5 | 5
Completed Cycle 1 | 2 | 6 | 3 | 1 | 3 | 2
Received Treatment (Number of subjects in each arm, who enrolled in study and received study treatment.) | 3 | 7 | 5 | 1 | 3 | 2
Completed | 3 | 7 | 5 | 1 | 3 | 2
Not Completed | 0 | 0 | 1 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 2
Not completed — Subject did not meet entry criteria | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of the 27 subjects enrolled, only 17 completed Cycle 1 of study treatment, and are therefor considered evaluable. 5 subjects withdrew or were taken off study prior to receiving study drug, 1 came off study due to disease progression, 3 were removed from the study, and 1 chose to withdraw prior to completing Cycle 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 DL1 | Phase 1 DL-1 | Phase 1 DL-1a | Phase 1 DL-1b | Phase 1 DL-1c | Phase 1 DL-1d | Total
Number analyzed (Participants) | 3 | 7 | 6 | 1 | 5 | 5 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 1 | 1 | 1 | 1 | 6
  >=65 years | 3 | 5 | 5 | 0 | 4 | 4 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 3 | 1 | 1 | 2 | 14
  Male | 1 | 2 | 3 | 0 | 4 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 3 | 7 | 6 | 1 | 4 | 4 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 00 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 2 | 0 | 4
  White | 3 | 5 | 6 | 1 | 3 | 4 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 7 | 6 | 1 | 5 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Safety of Birinapant (TL32711) in Subjects With Acute Myeloid Leukemia, Myelodysplastic Syndromes and Acute Lymphoblastic Leukemia. Acute Lymphocytic Leukemia.
Description: Safety of birinapant will be measured as the number of adverse events per dosing level occurring with greater than 5% frequency in the total evaluable subject population. Adverse events are any untoward medical occurrences experienced by research study participants. These events are documented and assessed for severity and relation to the study drug by the treating investigator, using the Common Terminology for Criteria for Adverse Events for severity, and information on known side effects of the study drug for relation.
Time Frame: First day of study treatment to 30 days after last study treatment. The average length of time for adverse event monitoring was 14 weeks.
Measure: Number; unit: Adverse Events
Arm/Group | Phase 1 DL1 | Phase 1 DL-1 | Phase 1 DL-1a | Phase 1 DL-1b | Phase 1 DL-1c | Phase 1 DL-1d
Number analyzed (Participants) | 3 | 7 | 5 | 1 | 3 | 2
Adverse Events | 25 | 34 | 35 | 10 | 3 | 2

2. Primary Outcome: Number of Dose Limiting Toxicities Per Dosing Level.
Description: This outcome measure will be defined as the number of dose limiting toxicities per dosing level. Dose limiting toxicities are pre-defined medical events that may be related to the dosing of the study drug. These toxicities are documented and assessed for severity based on pre-defined thresholds, and may result in modification of the study drug dosing.
Time Frame: as for outcome 1
Measure: Number; unit: Dose Limiting toxicities
Arm/Group | Phase 1 DL1 | Phase 1 DL-1 | Phase 1 DL-1a | Phase 1 DL-1b | Phase 1 DL-1c | Phase 1 DL-1d
Number analyzed (Participants) | 3 | 7 | 5 | 1 | 4 | 2
Dose Limiting toxicities | 2 | 0 | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Phase 1 DL1 vs Phase 1 DL-1 vs Phase 1 DL-1a vs Phase 1 DL-1b vs Phase 1 DL-1c vs Phase 1 DL-1d; Test type: Other; Based on the dose limiting toxicities occurring in each dosing cohort, a maximum tolerated dose (MTD) may be determined by assessing the highest dosing level presenting no dose limiting toxicities. An MTD of 17mg/m2 twice weekly was established

ADVERSE EVENTS:
Time Frame: Adverse events will be captured for each subject from the period from their initiation of study treatment to 30 days following their last administration of study treatment. The average length of time for adverse event monitoring was 14 weeks.
Description: Some adverse events were reported, assessed, and monitored per the CTCAE terminology using the Organ Class System rather than the specific event description. Ongoing adverse events have been captured as a single incidence to reflect the most severe grade of each event.
Groups:
- Phase 1 DL-1d: 22mg/m2/dose IV twice per week x 4weeks of 4 week cycle
  Birinapant: IV formulation to be given weekly 3 weeks out of 4 week cycle or 4 weeks our of a 4 week cycle as a 30 minute infusion
Arm/Group | Phase 1 DL1 | Phase 1 DL-1 | Phase 1 DL-1a | Phase 1 DL-1b | Phase 1 DL-1c | Phase 1 DL-1d
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/7 | 5/6 | 0/1 | 4/5 | 1/5
Serious Adverse Events (participants affected / at risk) | 3/3 | 6/7 | 5/6 | 1/1 | 4/5 | 3/5
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 5/6 | 1/1 | 4/5 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 DL1 (N=3) | Phase 1 DL-1 (N=7) | Phase 1 DL-1a (N=6) | Phase 1 DL-1b (N=1) | Phase 1 DL-1c (N=5) | Phase 1 DL-1d (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 1 (3) | 1 (1) | 2 (4) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0)
Serum amylase increase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Increase creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Bell's palsy
Peripheral motor neurpathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decrease neutrophil count (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection, bladder (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Sudden death NOS (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspena (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 DL1 (N=3) | Phase 1 DL-1 (N=7) | Phase 1 DL-1a (N=6) | Phase 1 DL-1b (N=1) | Phase 1 DL-1c (N=5) | Phase 1 DL-1d (N=5)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Disorders Other- Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Thrombocytopenia (Investigations) | 1 (1) | 7 (7) | 5 (5) | 1 (1) | 3 (3) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient Unilateral Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 5 (5) | 1 (1) | 3 (3) | 0 (0)
Neutropenia (Investigations) | 2 (2) | 7 (7) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flashing lights (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Leukopenia (Investigations) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, jaw sensitivity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio Myopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Watering Eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Scleral Hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth sores (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Petechiae
Mouth Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leg Pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Subcutaneous Disorders, Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — skin abnormalities which are wart-like in appearance
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection, Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Groin, Fungal
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gum Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and Urinary Disorders, Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Burning
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain, left trunk (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain, right trunk (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Herpes Zoster
Autoimmue disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
White Blood Cell Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — On neck
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain, back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Local Facial Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes